CLINICAL TRIAL: NCT04971473
Title: An Open, Single-arm, Self-controlled, Multi-center Phase 3 Study to Compare the Efficacy and Safety of rhTSH as An Adjunctive Diagnostic Tool in Differentiated Thyroid Cancer Patients Who Had Been Thyroidectomized Vs. Patients Who After Thyroid Hormone Withdrawal
Brief Title: Comparison of the Efficacy and Safety of rhTSH as An Adjunctive Diagnostic Tool in Differentiated Thyroid Cancer Patients Who Had Been Thyroidectomized Vs. Patients Who After Thyroid Hormone Withdrawal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGTSH004
Record Dates: First submitted 2021-07-07; First posted 2021-07-21 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-03

CONDITIONS: Differentiated Thyroid Cancer
MeSH Terms: interventions — Thyrotropin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rhTSH+Thyroid hormone withdrawal (Experimental): rhTSH: rhTSH(0.9 mg) was administered intramuscularly (IM) once daily (qd) for 2 days. Twenty-four hours following the second dose of rhTSH.Oral radioiodine was given 24 hours after the second injection of rhTSH, and scanning was done 48 hours after the radioiodine administration.
  Thyroid hormone withdrawal: Patients stop taking thyroid hormone for 14 days, and then monitor the level of thyroid stimulating hormone every week. When TSH>30mU/L, an ablative activity of 131I was administered.and scanning was done 48 hours after the radioiodine administration.
  Interventions: Biological: rhTSH

INTERVENTIONS:
Biological: rhTSH — Scanning was done 48 hours after the radioiodine administration. Each patient was scanned first following rhTSH and then scanned after thyroid hormone withdrawal.
  Other Names: recombinant human thyroid stimulating hormone

SUMMARY:
This is A non-blinded trial. Oral radioiodine was given 24 hours after the second injection of rhTSH, and scanning was done 48 hours after the radioiodine administration. Each patient was scanned first following rhTSH and then scanned after thyroid hormone withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily sign the informed consent form (ICF).
* Age 18-75 years old, either male or female.
* Patients with diagnosed differentiated papillary or follicular thyroid carcinoma, including papillary-follicular variant,.
* Patients with a total or near-total thyroidectomy within 6 weeks prior to administered.
* Low iodine diet for 4 weeks prior to randomized.

Exclusion Criteria:

* Pregnant or breast feeding women.
* Patients with other malignancies (exception for in situ cervix uterine cancer, baso cellular skin cancer or breast cancer in remission)
* Subjects who are unsuitable to the trial in combination with other serious diseases, as identified by the investigator.
* Subjects who have participated in another clinical trial of a new drug or medical instrument within 1 months before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
the rate of concordant scans | 48 hours after the radioiodine administration
  scan findings in agreement in a given patient using each preparation method

CONTACTS AND LOCATIONS:
Overall Officials: Yansong Lin, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lin Y, Wen Q, Fu W, Yang H, Gao Y, Li Z, Huang J, Gao Z, Wu J, Lv Z, Lu K, Chen Y, Yang A, OuYang W, Zhang S, Zhou H, Deng Z, Chen Z, Ding Y, Yuan C, Li L, Lin C, Sang S, Cheng Z, Cheng Y. RhTSH in aiding dynamic assessment in patients with differentiated thyroid Cancer. Eur J Nucl Med Mol Imaging. 2025 Dec;53(1):389-397. doi: 10.1007/s00259-025-07349-1. Epub 2025 Jun 9. PMID 40488858